CLINICAL TRIAL: NCT02058537
Title: Bethanechol for Treatment of Eosinophilic Esophagitis (EoE)
Brief Title: Bethanechol for Eosinophilic Esophagitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Initial PI left, study not continued
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Assouline-Dayan, Yehudith, Clinical Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bethanechol
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Bethanechol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bethanechol (Experimental): Oral administration of 25 milligrams of bethanechol taken twice daily for a minimum of 7 days. Total dose taken daily for a minimum of 7 days is 50 mg.
  Interventions: Drug: Bethanechol

INTERVENTIONS:
Drug: Bethanechol — Due to the fact that this study has only 1 arm and all study subjects will receive the study drug in the same manner and dose, there are no other details to cover.

SUMMARY:
The primary goals of this study are to ease the symptoms of patients with Eosinophilic Esophagitis (EoE) and to test the effectiveness of the drug bethanechol in relieving those symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 18-75
* Symptoms associated with EoE such as dysphagia, heartburn, vomiting, abdominal pain, food impaction
* Subject has signed informed consent for the administration of bethanechol that informs the patient of potential adverse events
* Clinically or pathologically proven EoE

Exclusion Criteria:

* Known allergy to bethanechol
* Asthma
* Pregnant or breast-feeding women
* Severe neurological problems
* Severe diabetes
* Achalasia
* Known allergy to lidocaine or other local anesthetic
* Hypothyroidism
* Peptic ulcer
* Pronounced bradycardia or hypotension
* Vasomotor instability
* Coronary artery disease
* Epilepsy
* Parkinsonism
* Weakened gastrointestinal or bladder wall
* Mechanical obstruction of the gastrointestinal tract or bladder neck
* Urinary bladder surgery in the 6 months prior to the study
* Gastrointestinal resection and anastomosis
* Spastic gastrointestinal disturbances
* Acute inflammatory lesions of the gastrointestinal tract
* Peritonitis
* Marked vagotonia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yehudith Assouline-Dayan, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bethanechol
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bethanechol
Number analyzed (Participants) | 3
Age, Categorical [Number; unit: participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.67 (16.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline High Resolution Esophageal Manometry With Impedance to Day 7
Description: The high resolution esophageal manometry with impedance involves a thin, pressure-sensitive tube that is passed through the nose and into the stomach. Once in place, the tube is pulled slowly back into the esophagus (food pipe). When the tube is in the esophagus, the patient is asked to swallow several times while swallowing water, applesauce, crackers, and marshmallows. These swallows will be completed while laying down, sitting upright, and standing. The pressure of the muscle contractions will be measured along several sections of the tube. The tube is removed after the tests are completed. This test allows for a quantitative measure of the pressure in the esophagus that can be correlated to difficulty or ease of bolus swallowing.
Time Frame: Day 1 and Day 7
Population: We did not do the data analysis since the originating PI left the institution and the study was terminated.
Arm/Group | Bethanechol
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline Evaluation of Esophageal Function Questionnaire to Day 7
Description: This questionnaire allows the patient to assess their own symptoms and report their opinions about drug effectiveness.
Time Frame: Day 1 and Day 7
Population: We did not do the data analysis since the originating PI left the institution and the study was terminated.
Arm/Group | Bethanechol
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Change From Baseline Composite Vital Signs to Day 7
Description: Vital signs include temperature, heart rate, breathing rate, and blood pressure. This variables will be measured during the study in order to assess any negative systemic effects of the study drug. These measurements are assessed as a composite and not individually therefore are grouped together as one outcome measure.
Time Frame: Day 1 and Day 7
Population: We did not do the data analysis since the originating PI left the institution and the study was terminated.
Arm/Group | Bethanechol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Bethanechol
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No